CLINICAL TRIAL: NCT03401658
Title: Feasibility Assessment of a Sensor Technology for Out-of-hospital Remote Surveillance of Surgical Site Infections
Brief Title: Early Detection of Surgical Wound Infections Using Sensor Technology
Acronym: SSI-Sensor
Status: Withdrawn | Type: Observational
Why Stopped: Funding stopped
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: 1175
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Surgical Wound Infection; Heart; Surgery, Heart, Functional Disturbance as Result
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Sensor light detector — The intervention is based on a sensor technology that gathers data and transmit it to another location for processing. The monitoring utilises an LED light source, an integral detector set which has variance from device to device and chromatic based algorithms for extraction of information from the detectors. The integration of these components into a system provides robustness and stability for operation. The availability of smartphones which possess high quality cameras and constant internet connectivity provides an ideal platform for multimedia clinical data collection and real-time patient-provider communication.

SUMMARY:
Infections that are caused by surgical incision are commonly known as surgical site infections (SSI). A surgical wound infection can develop at any time after surgery until the wound has healed (usually two to three weeks after the operation). Very occasionally, an infection can occur several months after an operation. About 5 in 100 patients develop SSI after hospital discharge. During the patient's stay in hospital, nurses routinely change their wound dressings to check for any signs of infection. However, since infections develop after patients leave hospital it is difficult for staff to monitor signs in patients' homes. In some hospitals, staff may contact patients in their homes to check on their wounds but most of the time it is not possible. The recent improvement in surgical operations means that more patients are discharged from hospital earlier than they would have been in the past even before their wounds are healed. Increasingly, patients develop SSI after leaving hospital particularly among the more vulnerable high risk groups. Signs of SSI may not always be recognised by the patient and delays in seeking care leads to serious infection-related complications. The investigators wish to fit a device onto the patients' personal mobile phone camera lens. This will allow patients to take pictures of their wound routinely at home submit images automatically to a computer at the hospital for analysis. Staff at the hospital will alert the patient if the results strongly that indicate signs of infection and an appropriate treatment plan put into place for you. This type of technology has never been used in this application before so, the investigators plan in this study to find out whether it can accurately detect early signs of wound infections and whether it is easy to use, acceptable to the patient and their health care professionals. A total of 40 patients will be invited to take part in the study over a period of 12 months.

DETAILED DESCRIPTION:
BACKGROUND:

Surgical site infections (SSI) are notable common complications of cardiothoracic surgery and frequently results in readmission and diminished quality of life. SSI may range from a simple spontaneous limited wound discharge to the more severe deep-seated sternal infections. These combined account for about 16% of all hospital acquired infections with an estimated doubling effect on postoperative length of hospital stay and cost of care. The high costs associated with SSI arise primarily because of prolonged hospital stays and the need for repeated surgical procedures in these patients. Patients with chronic obstructive pulmonary disease (COPD), smoking, diabetes, malnutrition, obesity and need for bilateral harvest of the internal thoracic artery during surgery have been identified as having significantly higher risk of infections. Socio-economic factors are also known contributors to SSI.

Many specialist cardiothoracic centres in the UK have internal governance structures within the hospital to monitor the outcomes of its procedures each year to ensure that the work done is of the highest quality and keeps patients safe. However one area of greatest concern is the apparent lack of robust measures for out-of-hospital wound management for patients that have undergone surgical procedures. With shorter hospitalisations due to improved surgical techniques, patients are often discharged from hospital before their wounds are fully healed. Recent studies suggest that inadequate post-discharge communication and untimely, infrequent follow-up contribute to poorer outcomes (e.g. readmission).

The absence of robust systems for SSI surveillance and monitoring of wound healing after hospital discharge presents a big challenge and often results in serious consequences. Some patients are more vulnerable to surgical site infections particularly after hospital discharge. Consequently wound infections become deep-seated and problematic to treat within the primary care setting. Several reasons are known to contribute to susceptibility to surgical wound infections with the international literature reporting that deprivation is a significant risk factor. Evidence also shows that some patients are unable to self-diagnose their wound infections because of lack of sufficient knowledge at the point of hospital discharge. It is also known that some patients find it hard to access GP services due to lack of the availability for urgent appointments. Having to wait to see a GP is often a barrier to seeking help. Others may be unable to contact their GP practices due to increasing demand.

Evidence from our hospital indicates that from September 2014 to August 2016, there was a combined in-hospital surgical site infection rates for sternal and graft harvest sites of 6.3% (172 out of 2711) for patients that had undergone coronary artery bypass graft surgery alone. In addition, about 1% (27 out of 2711) of these patients had severe deep-seated surgical site infections after hospital discharge that required hospital readmission and additional extensive utilisation of NHS resources for their care. Even if the numbers are understated, surgical site infection represents significant costs to the NHS, ranging from £2,100 to £10,500 per infection depending on the nature of the surgery. Expert opinion suggests that costs can be as high as £20,000 per surgical site infection for complex surgery and up to £14,000 for the more general surgery.

This feasibility project will address this concern through the development and optimisation of an early warning sensor-based technology for remote monitoring of out-of-hospital surgical site wound infections. In addition, the project will explore issues associated with the remote application of the sensor technology itself and develop measures to address them.

RATIONALE, AIMS AND OBJECTIVES OF THE RESEARCH A significant number of patients are re-admitted into hospital after cardiac surgery under the emergency care pathway because of severe surgical site infections. These complications occur because patients are not adequately monitored once they are discharged from hospital and often they do not alert their GP until the infection site becomes deep seated (inside tissues and bones). This is due to their inability to tell the difference between inflammation and early signs of superficial infections that could easily be treated by their GP. Treatment of deep-seated infection requires hospitalisation and costs the NHS in excess of £700 million annually.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they had a planned or urgent elective coronary artery bypass graft surgery, 18 years or older, with high risk factors such as elderly patients (≥75 years old) living alone, having morbid obesity (BMI>37 kg/m2), diabetes, COPD, are smokers or have a planned bilateral harvest of the internal thoracic artery.

Exclusion Criteria:

* Patients will be excluded if they are: undergoing additional procedures such as antimicrobial-impregnated incision drapes; have existing wound dressing prior to discharge, undergoing chemotherapy, immunosuppressive therapy or steroids; use of antibiotics for an active infection; therapeutic radiation or renal dialysis; intra-aortic balloon pump or mechanical assist device preoperatively. They will be excluded if they have an abnormal skin condition around the surgical incision site; have neutropenia, have HIV infection with CD4 count <350 per mm3; have sensitivity or allergic to cyanoacrylate, isopropyl alcohol, iodine, iodine-containing products or tape.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients identified from the surgical waiting or operation list. Patients should be resident within the Liverpool area and must be smartphone users. The mobile phone must have the facility to be locked by either a code or fingerprint recognition. Only high-risk patients that meet the inclusion criteria will be approached for consent, by the consultant performing the initial assessment before the procedure or the research nurse, either in the pre admission clinic or in hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Number of surgical site infections that can reliably be detected using the sensor technology | Daily for 30 days
  Number of surgical sites infections detected

SECONDARY OUTCOMES:
Proportion of patients that find the sensor technology acceptable | Questionnaire administered once at day 30
  Acceptability and easy of application by patients

CONTACTS AND LOCATIONS:
Overall Officials: Mark Field, MBBS, PhD, Principal Investigator — Liverpool Heart & Chest Hospital
Locations (1):
- Liverpool Heart and Chest Hospital, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Background] Gibson A, Tevis S, Kennedy G. Readmission after delayed diagnosis of surgical site infection: a focus on prevention using the American College of Surgeons National Surgical Quality Improvement Program. Am J Surg. 2014 Jun;207(6):832-9. doi: 10.1016/j.amjsurg.2013.05.017. Epub 2013 Oct 10. PMID 24119885
- [Background] Perencevich EN, Sands KE, Cosgrove SE, Guadagnoli E, Meara E, Platt R. Health and economic impact of surgical site infections diagnosed after hospital discharge. Emerg Infect Dis. 2003 Feb;9(2):196-203. doi: 10.3201/eid0902.020232. PMID 12603990
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699